CLINICAL TRIAL: NCT04399317
Title: Flow Controlled Ventilation in ARDS Associated With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: MRC-05-018
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-05

CONDITIONS: ARDS Associated With COVID-19
Keywords: ARDS; COVID-19; Ventilation
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: randomization to treatment or control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the technical facts (use of a different mechanical ventilator) only the participants (who are sedated) and the outcome assessor will be blinded for the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): This is the treatment group. Patients will be ventilated using the new device (Evone) applying flow controlled ventilation for 48 hours. Ventilation parameters will be assessed every 6-8 hours. All other treatment will be unchanged and according to institutional standards.
  Interventions: Device: Flow controlled ventilation (Evone-ventilator)
- Group B (No Intervention): These patients will be treated according to institutional standards. Only data will be collected. This is the control group.

INTERVENTIONS:
Device: Flow controlled ventilation (Evone-ventilator) — The new ventilation technique will be applied
  Arms: Group A

SUMMARY:
The pandemic of a newly upcoming viral disease which is associated with COVID-19 puts the whole world's health system under pressure.

Patients suffering from this disease mainly develop respiratory symptoms, which can lead to severe acute respiratory distress syndrome (ARDS) necessitating ICU, admission in 10-20% of the cases admitted to hospital. In addition to these symptoms, patients show lymphopenia, cardiac symptoms and altered coagulation profiles. Although those patients are treated in the ICU the mortality is up to 20% due to multiorgan failure. The aim of this study is to show non-inferiority of flow-controlled ventilation compared to standard (lung protective ventilation).

Methods:

After admission to the ICU, the patients will receive information about the study and informed consent will be taken. Upon reaching the criteria for moderate to severe ARDS (P/F ratio below 200 mmHg and PEEP above 5 cmH2O) the patients will be randomized. In the treatment group (group A) the ultra-thin ventilation tube will be placed through the existing tube. Then flow-controlled ventilation will be applied for 48 hours. In the other group (group B) ventilation will be performed according to the lung protective strategy. All other treatment will be unchanged.

Data-collection will be started 1 hour after initiation of the study. Primary end point is PaO2.

DETAILED DESCRIPTION:
The pandemic of a newly upcoming viral disease which is associated with COVID-19 puts the whole world's health system under pressure.

Patients suffering from this disease mainly develop respiratory symptoms, which can lead to severe acute respiratory distress syndrome (ARDS) necessitating ICU admission in 10-20% of the cases admitted to hospital. In addition to these symptoms, patients show lymphopenia, cardiac symptoms and altered coagulation profiles. Although those patients are treated in the ICU the mortality there is up to 20% due to multiorgan failure. Currently, there is no proven therapeutic strategy next to symptomatic treatment.

Although the severely ill patients will need intubation and invasive ventilation according to ARDS treatment strategies including low tidal volumes and low end-expiratory pressures, not all patients recover their pulmonary function.

Flow control ventilation (FCV) is a recently developed ventilation strategy which allows to keep the intrapulmonary pressures low while achieving optimal gas exchange. It had been proven in animal models to improve pulmonary function and oxygenation and in cases with ARDS.

Flow Controlled Ventilation mode is a unique ventilation technique in which inspiration as well as expiration are controlled i.e. actively performed. This is achieved by generating a continuous flow into the patient's lungs during inspiration or a continuous (negative) flow, sucking gasses out of the patient's lungs.

The continuous flow without ventilation pauses, results in linear increases and decreases in intratracheal pressures. As a result, the mean airway pressure will be higher compared to conventional large bore Volume Controlled Ventilation or Pressure Controlled Ventilation (PCV). Therefore, the bronchiole and alveoli will be kept open during ventilation facilitating oxygen uptake to the blood. Moreover, the continuous gas flow enhances gas mixture in the lungs also improving gas exchange. Altogether, FCV results in more efficient ventilation as compared to conventional ventilation techniques.

Evone® is the only commercially available ventilator applying FCV ventilation mode, thus directing the inspiration as well as the expiration. Evone's FCV® ventilation mode is based on a controlled inspiration and expiration flow from a set PEEP to a set peak pressure and vice versa. The inspiratory flow is continuously controlled by advanced mass flow regulators; the expiratory flow is controlled by regulated suctioning.

Aim of the study This study aims to demonstrate the positive effects on oxygenation of flow-controlled ventilation compared to conventionally ventilated patients (pressure control ventilation) in patients suffering from ARDS associated with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with ARDS due to COVID-19
* need for mechanical ventilation
* P/F ratio <200mmHg
* PEEP of at least >5cmH2O
* BMI less 30 kg/ m2

Exclusion Criteria:

* Refuse to sign the consent
* Chronic Respiratory disease
* Acute or chronic Cardiovascular disease
* Pregnancy
* Already under special therapy (prone position and/or ECMO)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
arterial oxygen partial pressure (PaO2) | during 48 hours of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lance, MD, PhD, Principal Investigator — Hamad Medical Corporation, Weill-Cornell-Medicine Qatar, Qatar University
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding sharing information will be taken at later stage.

REFERENCES:
- [Derived] Roehrig S, Ait Hssain A, Shallik NAH, Elsaid IMA, Mustafa SF, Smain OAM, Molokhia AA, Lance MD. Flow controlled ventilation in Acute Respiratory Distress Syndrome associated with COVID-19: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Sep 11;21(1):781. doi: 10.1186/s13063-020-04708-1. PMID 32917259